CLINICAL TRIAL: NCT06748521
Title: Efficacy and Safety of Dynamic CtDNA-guided Targeted Therapy in Patients with Previously Untreated Diffuse Large B-cell Lymphoma
Brief Title: Dynamic CtDNA-guided Targeted Therapy in DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0511200
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: R-CHOP + X

INTERVENTIONS:
Drug: R-CHOP + X — Eligible participants will receive 1 cycle of R-CHOP therapy with genotyping and ctDNA testing at C1D14. Chemotherapy sensitive patients with C1D14 ctDNA negative or ctDNA LFC ≥ 2 will continue to receive R-CHOP therapy for up to 6 courses. Potentially resistant patients with C1D14 ctDNA positive and LFC < 2 were stratified by DLBCL genotyping and treated with cycle 2-6 R-CHOP in combination with obutinib or decitabine or lenalidomide or Chidamide.

SUMMARY:
This is a prospective, single-arm, noninferiority trial involving patients with previously untreated CD20-positive DLBCL. The aim of this study is to determine the efficacy and safety of treatment stratified based on ctDNA dynamic changes after one cycle of chemotherapy and the targeted therapy based on DLBCL genotype.

A total of 108 patients were planned to be enrolled in this trial, and the patients were stratified according to the dynamic changes of ctDNA after one cycle of chemotherapy: the chemotherapy-sensitive group continued the original R-CHOP regimen, and the potential drug resistance group received genotype-guided targeted drug combination. The whole trial included a screening period (day -28 to day -1), a treatment period, and a 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age 18-75 years at the time of signing Informed Consent Form and willingness to comply with study protocol procedures
* Previously untreated participants with CD20-positive DLBCL
* IPI score 2-5
* ECOG Performance Status of 0, 1, or 2
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Contraindication to any of the individual components of R-CHOP or Obutinib or Decitabine or Lenalidomide or Chidamide
* Have received systemic or local treatment including chemotherapy in the past
* Have received autologous stem cell transplantation in the past
* Past medical history of other malignant tumors, except basal cell carcinoma of the skin and cervical cancer in situ
* Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulopathy, connective tissue diseases, severe infectious diseases and other diseases
* Primary central nervous system lymphoma
* Left ventricular ejection fraction ≦50%
* Other concurrent and uncontrolled situation which will affect the patient's medical status based on researchers' decision
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma):

  * ANC < 1.0 x 10^9/L
  * PLT < 75 x 10^9/L
  * Hb < 100g/L
  * Serum AST and ALT ≥ 2.5 x ULN
  * Total bilirubin ≥ 1.5 x ULN
  * Serum creatinine ≥ 1.5 x ULN
* Psychiatric patients or other patients who are known or suspected to be unable to fully accomplish with the research protocol
* Pregnant or lactating women
* Patients with positive HbsAg test results need to undergo HBV-DNA test and can be admitted to the group after turning negative. In addition, if the HBsAg test result is negative, but the HBcAb test is positive (regardless of the HBsAb status), HBV-DNA is also required；if the result is positive, patients also need to be treated to become negative before entering the group
* Patients living with HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-12-13 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | End of Cycle 6 (each cycle is 21 days)
  CR rate at the end of treatment. Defined as the proportion of participants who achieved CR at the end of treatment.

SECONDARY OUTCOMES:
2-year progression-free survival (PFS) rate | 2 years
  PFS, defined as the time from enrollment to the first occurrence of disease progression or relapse using the 2014 Lugano Response Criteria or death due to any cause, whichever occurs first; as determined by the investigator. The 2-year PFS rate was the percentage of patients who did not experience disease progression or death within two years of enrollment.
2-year Overall survival (OS) rate | 2 years
  OS defined as the time from enrollment to death from any cause. The 2-year OS rate was the percentage of patients who did not die within two years of enrollment.
The incidence and severity of adverse events were determined according to the NCI CTCAE v5.0 rating scale | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

IPD SHARING:
Plan to Share IPD: No